CLINICAL TRIAL: NCT01906008
Title: Phase II, Randomized, Placebo-Controlled Study of Minocycline for Reducing Symptom Burden in Patients With Colorectal Cancer
Brief Title: Phase II Study of Minocycline for Reducing Symptom Burden in Colorectal Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0323; NCI-2014-01291 (Registry Identifier: NCI CTRP); RSG-13-241-01-PCSM (Other: Amercian Cancer Society)
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; CRC; Acute peripheral neuropathy; Numbness; Pain; Loss of motor function; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn; Placebo; Questionnaires; Surveys; Sensory tests
MeSH Terms: conditions — Colorectal Neoplasms; Hypesthesia; Pain; cyclopia sequence | interventions — Minocycline; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Minocycline (Experimental): Group 2 receives minocycline 200 mg orally for the first dose, then 100 mg orally every 12 hours for 4 months beginning at chemotherapy initiation. Completion of questionnaires at baseline, 1 time each week, at each chemo cycle, at end of treatment visit, and at 6 month follow up visit. Sensory test performed at baseline, 2 months, end of treatment visit, and at 6 month follow up visit.
  Interventions: Drug: Minocycline; Behavioral: Questionnaires; Behavioral: Sensory Test
- Placebo (Placebo Comparator): Group 1 receives a placebo 200 mg orally for the first day of chemotherapy, then 100 mg doses every 12 hours for 4 months beginning at chemotherapy initiation. Completion of questionnaires at baseline, 1 time each week, at each chemo cycle, at end of treatment visit, and at 6 month follow up visit. Sensory test performed at baseline, 2 months, end of treatment visit, and at 6 month follow up visit.
  Interventions: Drug: Placebo; Behavioral: Questionnaires; Behavioral: Sensory Test

INTERVENTIONS:
Drug: Minocycline — 200 mg by mouth for the first dose, then 100 mg by mouth every 12 hours for 4 months beginning at chemotherapy initiation.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Minocycline
Drug: Placebo — 1 placebo by mouth for the first day of chemotherapy, then 1 dose every 12 hours for 4 months beginning at chemotherapy initiation.
  Arms: Placebo
Behavioral: Questionnaires — Completion of questionnaires at baseline, 1 time each week, at each chemo cycle, at end of treatment visit, and at 6 month follow up visit.
  Other Names: Surveys
Behavioral: Sensory Test — Sensory test performed at baseline, 2 months, end of treatment visit, and at 6 month follow up visit.

SUMMARY:
The goal of this clinical research study is to learn if minocycline can reduce numbness, pain, and/or loss of motor function in patients with colorectal cancer. In this study, minocycline will be compared to a placebo.

The study doctor can explain how the study drug is designed to work.

A placebo is not a drug. It looks like the study drug, but it is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Nearly 40% of patients with colorectal cancer who receive oxaliplatin-based chemotherapy experience neuropathy (nerve damage that can include numbness, pain, and/or loss of motor function). Sometimes, this nerve damage is serious enough that the chemotherapy dose has to be lowered or stopped completely. Researchers want to find out if taking minocycline can lower the side effects caused by chemotherapy given to treat colorectal cancer.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being in either group:

* If you are in Group 1, you will take a placebo.
* If you are in Group 2, you will take minocycline.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

Starting on Day 1 of Cycle 1 of chemotherapy, you will start taking the study drug/placebo capsule by mouth, twice a day every day.

You should take the study drug/placebo with a full glass (8 ounces) of water. You may take it with or without food, but if it causes an upset stomach, you should take it with food.

You should not lie down for at least 30 minutes after taking the study drug/placebo to reduce the risk of side effects.

Study Visits:

Before you start taking the study drug/placebo:

* You will complete 4 questionnaires about pain and other symptoms, and your quality of life. You will also complete a questionnaire about your tobacco history. It should take about 15-25 minutes to complete all questionnaires.
* You may complete a sensory test. For this test, researchers will try to find out how sensitive you are to touching things such as small bumps on a board. This test will take about 10 minutes to complete.
* If possible, blood (about 6 teaspoons) will be drawn to test for markers of inflammation. Markers of inflammation are found in the blood and may be related to your symptoms.

  1 time each week:
* You will complete a questionnaire in the clinic or by telephone about any symptoms you may be having and how they may be affecting your daily activities. The questionnaire should take about 3-5 minutes to complete each time.

At each chemotherapy cycle:

* You will fill out 2 questionnaires in the clinic or by telephone about pain and other symptoms. It should take about 10-15 minutes to complete the questionnaires.
* The study staff will make a count of the number of pills that you took so far. If you are coming to the MD Anderson or Harris Health clinic, bring the study drug/placebo container (along with any remaining drug/placebo).

At about 2 months:

* If you return to the MD Anderson or Harris Health clinic for this visit, the following additional procedures will be performed:
* If possible, blood (about 6 teaspoons) will be drawn to test for markers of inflammation.

You may complete a sensory test. This test will take about 10 minutes to complete.

End-of-Treatment Visit (at about 4 months):

* You will fill out the 4 questionnaires in the clinic or by telephone about your symptoms. It should take about 15-20 minutes to complete all of the questionnaires.
* The study staff will make a count of the number of pills that you took so far.

If you return to the MD Anderson or Harris Health clinic for this visit:

* If possible, blood (about 6 teaspoons) will be drawn to test for markers of inflammation.
* You may complete a sensory test. This test will take about 10 minutes to complete.
* You must bring the study drug/placebo container (along with any remaining drug/placebo).

Length of Study:

You may continue taking the study drug/placebo for up to 4 months, if there are no treatment delays. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation in the study will be over at the End-of-Study visit.

End-of-Study Visit:

At about 6 months, the following tests and procedures will be performed:

°You will fill out 4 questionnaires in the clinic or by telephone about pain and other symptoms and your quality of life. You will also complete a questionnaire about your tobacco history. It should take about 15-25 minutes to complete all of the questionnaires.

If you return to the MD Anderson or Harris Health clinic for this visit:

* If possible, blood (about 6 teaspoons) will be drawn to test for markers of inflammation.
* You may complete a sensory test. This test will take about 10 minutes to complete.

This is an investigational study. Minocycline is FDA approved and commercially available for the treatment of bacterial infection. Its use in this study is investigational.

Up to 166 participants will be enrolled in this study. Up to 83 will be enrolled at the Harris Health System.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathologically proven diagnosis of CRC seen either at MD Anderson or LBJ.
2. Patients > or = 18 years old.
3. Patients who qualify for oxaliplatin-based chemotherapy (in the adjuvant or metastatic setting) and are likely to receive at least 3 months of oxaliplatin.
4. Patients who speak English or Spanish (due to language options for the MDASI version being used in this study, we are only recruiting English-speaking or Spanish-speaking patients).
5. Patients with an NCI-CTCv4 sensory neuropathy score of 0.
6. Patients with adequate renal function (serum creatinine must be < 1.5 times the upper limit of the institutional normal range) and no prior renal disease that in the opinion of the attending physician would make the patient ineligible to receive the study drug . Test results must be no more than 3 months old.
7. Patients with adequate hepatic function (total bilirubin must be < 2.0 times the upper limit of the institutional normal range; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be < 3.0 times the upper limit of the institutional normal range). Test results must be no more than 3 months old.
8. Patients willing and able to review, understand, and provide written consent.

Exclusion Criteria:

1. Patients continuously taking any minocycline within the last 15 days. Patients who have conditions that potentially preclude use of minocycline as determined by the treating physician.
2. Patients continuously taking systemic steroids within the last 15 days.
3. Patients with autoimmune disorders (for example, systemic lupus erythematosus or rheumatoid arthritis), who have been treated in the last 3 years.
4. Patients who are pregnant; the absence of pregnancy will be confirmed by negative urine test.
5. Hypersensitivity to any tetracyclines, or a history of other allergies or drug reactions that in the treating physician's judgment make the patient inappropriate for this study.
6. Patients receiving vitamin K antagonist (warfarin).
7. Patients with a BMI >40 (Obese Class III criteria).
8. Patients who will receive cetuximab or other targeted therapy where physicians may use topical doxycycline to reduce the rash associated with therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Eng, MD, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - LBJ Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 25, 2013 to May, 25 2017. Recruitment done at the University of Texas MD Anderson Cancer and LBJ.
Pre-assignment Details: Of the 122 participants enrolled 2 participant were excluded from the study before asssigment to groups.
Groups:
- Minocycline: Minocycline 100 mg twice a day during 4 months
- Placebo: Placebo 100 mg twice a day during 4 months
Period: Overall Study
Arm/Group | Minocycline | Placebo
Started | 59 | 61
Completed | 32 | 34
Not Completed | 27 | 27
Not completed — Lost to Follow-up | 2 | 0
Not completed — Oxaliplatin toxicity | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Did not start study med | 3 | 4
Not completed — Oxaliplatin stops | 10 | 8
Not completed — Hospice | 1 | 0
Not completed — Physician Decision | 3 | 3
Not completed — Lack of compliance of study med | 5 | 3
Not completed — Adverse Event | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 32 | 59
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (10.1) | 51.4 (10.1) | 52.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 22 | 41
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 6 | 12
  White | 23 | 26 | 49
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Average Area Under the Curve (AUC) for Numbness/Tingling Over 4 Months
Description: AUC for MDASI-numbness/tingling . Each item is rated on a 0 to 10 scale with 0 = symptom not present or no interference and 10 meaning the symptom severity is as bad as can be imagine or complete interference. For this study, the sub scale is the average of the 2 preselected items namely, numbness/tingling and fatigue. This subscale ranges from 0 to 10. The primary outcome is the average of the 120 -day area (4 months) under the curve for the sub scale. AUC ranges from 0 (0*120) to 1200 (10*120). To put this into perspective, the average AUC of 103.5 can also be thought of as an average daily AUC of 0.86 ( 103.5/120) on a 0 to 10 scale over the 120-day study period. Lower values represent better outcome while higher values represent worse outcome.
Time Frame: Baseline to 4 months
Measure: Mean (Standard Deviation); unit: Units on a scale *days
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 32 | 34
Units on a scale *days | 35.4 (27.35) | 31.5 (27.8)

2. Secondary Outcome: Average Area Under the Curve (AUC) for Fatigue Over 4 Months
Description: AUC for MDASI-fatigue . Each item is rated on a 0 to 10 scale with 0 = symptom not present or no interference and 10 meaning the symptom severity is as bad as can be imagine or complete interference. For this study, the sub scale is the average of the 2 preselected items namely, numbness/tingling and fatigue. This subscale ranges from 0 to 10. The primary outcome is the average of the 120 -day area (4 months) under the curve for the sub scale. AUC ranges from 0 (0*120) to 1200 (10*120). To put this into perspective, the average AUC of 103.5 can also be thought of as an average daily AUC of 0.86 ( 103.5/120) on a 0 to 10 scale over the 120-day study period. Lower values represent better outcome while higher values represent worse outcome.
Time Frame: Baseline to 4 months
Measure: Mean (Standard Deviation); unit: Units on a scale *days
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 32 | 34
Units on a scale *days | 47.92 (36.42) | 40.31 (30.92)

ADVERSE EVENTS:
Time Frame: The adverse events were monitoring/assessed from the first dose of study medication, up to 30 days after the last dose.
Arm/Group | Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 2/32 | 2/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline (N=32) | Placebo (N=34)
Hiperpigmentation spots (Skin and subcutaneous tissue disorders) | 1 | 0
Elevated LFT's (Metabolism and nutrition disorders) | 1 | 0
Elevated ALT (Metabolism and nutrition disorders) | 0 | 1
Elevated total Bilirrubin (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT01906008/Prot_SAP_000.pdf